CLINICAL TRIAL: NCT06852235
Title: Characteristics and Treatment Outcome of Liver Abscesses: An Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marco Magdy Wadie, Resident at Police Hospital, Assiut University
Other Study IDs: Liver abscess
Record Dates: First submitted 2025-02-22; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Liver Abscess
MeSH Terms: conditions — Liver Abscess

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To assess the frequency, clinical presentation, microbiological and radiological characteristics of liver abscesses.
2. To evaluate the management plan and treatment outcome of liver abscess.
3. To study risk factors of liver abscess.

DETAILED DESCRIPTION:
There is a paucity of information on liver abscesses' epidemiology and characteristics in the Middle East in general and Egypt in particular.

The incidence of liver abscess varies from one country to another. The annual incidence of pyogenic liver abscess has been estimated at 2.3 cases per 100,000 populations and 18-20 per 100 000 hospital admissions (Mohsen et al 2002, Kaplan et al 2004).

Liver abscess is a potentially life-threatening condition (Ahmed et al., 2016).

A review by Chan KS et al. of 16 pyogenic LA (PLA) articles showed mortality rates ranging from 0% to 15.7 % (Chan et al., 2022).

The etiology of LA can be bacterial (most often polymicrobial), parasitic (amebic essentially), mixed (pyogenic superinfection of parasitic abscess) or more rarely fungal (Nakanishi et al., 2009).

Microbes can invade the liver parenchyma by way of the bile ducts, blood stream (hematogenic, most often portal), or by contiguous spread, especially via the gallbladder bed (Yoo et al., 1993, Thomsen et al., 2007).

Advanced age, diabetes mellitus (DM) and the presence of underlying malignancy are considered major risk factors, and the latter is associated with a worse prognosis (Yoo et al., 1993, Thomsen et al., 2007).

The number of cryptogenic liver abscess cases has been on the rise, and no predisposing conditions (cryptogenic) was reported in 18% (McNeil et al. 2020).

The diagnosis of LA relies essentially on imaging. Sonography and CT scan lead to diagnosis in more than 90% of cases (Halvorsen et al., 1984).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of LA will be based on typical appearance on ultrasound (US) or computed tomography (CT) of abdomen with clinical features consistent with the diagnosis (fever, chills, jaundice, right upper quadrant pain/epigastric discomfort).
* US or CT-guided aspiration of pus from a hepatic lesion.
* Complete resolution of radiological abnormalities following antimicrobial therapy.

Exclusion Criteria:

* Liver abscess that occurs secondary to hydatid cyst.
* Liver abscess associated with underlying malignancy.
* Patient with incomplete medical records.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with liver abscess according to inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
1. To assess the frequency, clinical picture, microbiological and radiological characteristics of liver abscesses. | Baseline
  Data will be statistically evaluated by SPSS version 22. Numerical data will be expressed as means ± SDs.
  Categorical data will be expressed as frequencies (percentages).
  Comparison between groups will be conducted using t-test or Chi square test as appropriate.
  P value <0.05 will be considered as significant.

SECONDARY OUTCOMES:
2. To evaluate the management plan and treatment outcome of liver abscess. | Baseline
  Data will be statistically evaluated by SPSS version 22. Numerical data will be expressed as means ± SDs.
  Categorical data will be expressed as frequencies (percentages).
  Comparison between groups will be conducted using t-test or Chi square test as appropriate.
  P value <0.05 will be considered as significant.
3. To study risk factors of liver abscess. | Baseline
  Data will be statistically evaluated by SPSS version 22. Numerical data will be expressed as means ± SDs.
  Categorical data will be expressed as frequencies (percentages).
  Comparison between groups will be conducted using t-test or Chi square test as appropriate.
  P value <0.05 will be considered as significant.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Mahmoud Othman, doctorate, Study Director — Assiut University; Haidi Karam-Allah Ramadan, doctorate, Study Director — Assiut University

REFERENCES:
- [Background] Ahmed S, Chia CL, Junnarkar SP, Woon W, Shelat VG. Percutaneous drainage for giant pyogenic liver abscess--is it safe and sufficient? Am J Surg. 2016 Jan;211(1):95-101. doi: 10.1016/j.amjsurg.2015.03.002. Epub 2015 May 7. PMID 26033361
- [Background] Alkofer B, Dufay C, Parienti JJ, Lepennec V, Dargere S, Chiche L. Are pyogenic liver abscesses still a surgical concern? A Western experience. HPB Surg. 2012;2012:316013. doi: 10.1155/2012/316013. Epub 2012 Feb 19. PMID 22536008
- [Background] Baban FA. Clinical characteristic of amoebic liver abscesses in the North of Iraq. Saudi Med J. 2000 Jun;21(6):545-9. PMID 11500703
- [Background] Ballas ZK, Uthman SM. Amebic liver abscess in Lebanon. A report of 37 cases and a review of the literature. Am J Proctol. 1973 Jun;24(3):228-36. No abstract available. PMID 4707978
- [Background] Chan KS, Chia CTW, Shelat VG. Demographics, Radiological Findings, and Clinical Outcomes of Klebsiella pneumonia vs. Non-Klebsiella pneumoniae Pyogenic Liver Abscess: A Systematic Review and Meta-Analysis with Trial Sequential Analysis. Pathogens. 2022 Aug 26;11(9):976. doi: 10.3390/pathogens11090976. PMID 36145408
- [Background] Chiche L, Dargere S, Le Pennec V, Dufay C, Alkofer B. [Pyogenic-liver abscess: diagnosis and management]. Gastroenterol Clin Biol. 2008 Dec;32(12):1077-91. doi: 10.1016/j.gcb.2008.09.019. Epub 2008 Nov 18. French. PMID 19019604
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Background] Halvorsen RA, Korobkin M, Foster WL, Silverman PM, Thompson WM. The variable CT appearance of hepatic abscesses. AJR Am J Roentgenol. 1984 May;142(5):941-6. doi: 10.2214/ajr.142.5.941. PMID 6372412
- [Background] Huang CJ, Pitt HA, Lipsett PA, Osterman FA Jr, Lillemoe KD, Cameron JL, Zuidema GD. Pyogenic hepatic abscess. Changing trends over 42 years. Ann Surg. 1996 May;223(5):600-7; discussion 607-9. doi: 10.1097/00000658-199605000-00016. PMID 8651751
- [Background] Kaplan GG, Gregson DB, Laupland KB. Population-based study of the epidemiology of and the risk factors for pyogenic liver abscess. Clin Gastroenterol Hepatol. 2004 Nov;2(11):1032-8. doi: 10.1016/s1542-3565(04)00459-8. PMID 15551257
- [Background] Liu L, Chen W, Lu X, Zhang K, Zhu C. Pyogenic Liver Abscess: A Retrospective Study of 105 Cases in an Emergency Department from East China. J Emerg Med. 2017 Apr;52(4):409-416. doi: 10.1016/j.jemermed.2016.09.026. Epub 2016 Oct 17. PMID 27765437
- [Background] McNeil T, Daniel S, Gordon DL. Management of pyogenic liver abscess: a South Australian experience. ANZ J Surg. 2020 Nov;90(11):2274-2278. doi: 10.1111/ans.15963. Epub 2020 May 26. PMID 32455495
- [Background] Mohsen AH, Green ST, Read RC, McKendrick MW. Liver abscess in adults: ten years experience in a UK centre. QJM. 2002 Dec;95(12):797-802. doi: 10.1093/qjmed/95.12.797. PMID 12454322
- [Background] Mousa H, Al-Bluwi GSM, Al Drini ZFM, Gasmelseed HI, Alkoteesh JA, Babiker ZOE. Importation of Entamoeba histolytica and predominance of Klebsiella pneumoniae in liver abscesses: a 7-year retrospective cohort study from the United Arab Emirates. Trop Dis Travel Med Vaccines. 2021 Jun 12;7(1):17. doi: 10.1186/s40794-021-00140-8. PMID 34118991
- [Background] Mucke MM, Kessel J, Mucke VT, Schwarzkopf K, Hogardt M, Stephan C, Zeuzem S, Kempf VAJ, Lange CM. The role of Enterococcus spp. and multidrug-resistant bacteria causing pyogenic liver abscesses. BMC Infect Dis. 2017 Jun 26;17(1):450. doi: 10.1186/s12879-017-2543-1. PMID 28651522
- [Background] Nakanishi Y, Kayahara T, Yamashita Y, Okuno M, Nakamura F, Taniguchi Y, Inoue N, Nakatani Y, Hatamaru K, Shimizu T, Tanaka A, Yoshioka T, Seta T, Urai S, Uenoyama Y. [A case of ruptured giant liver cyst complicated by Candida infection]. Nihon Shokakibyo Gakkai Zasshi. 2009 Jul;106(7):1056-62. Japanese. PMID 19578314
- [Background] Solomkin JS, Mazuski JE, Bradley JS, Rodvold KA, Goldstein EJ, Baron EJ, O'Neill PJ, Chow AW, Dellinger EP, Eachempati SR, Gorbach S, Hilfiker M, May AK, Nathens AB, Sawyer RG, Bartlett JG. Diagnosis and management of complicated intra-abdominal infection in adults and children: guidelines by the Surgical Infection Society and the Infectious Diseases Society of America. Surg Infect (Larchmt). 2010 Feb;11(1):79-109. doi: 10.1089/sur.2009.9930. PMID 20163262
- [Background] Thomsen RW, Jepsen P, Sorensen HT. Diabetes mellitus and pyogenic liver abscess: risk and prognosis. Clin Infect Dis. 2007 May 1;44(9):1194-201. doi: 10.1086/513201. Epub 2007 Mar 28. PMID 17407038
- [Background] Yoo HM, Kim WH, Shin SK, Chun WH, Kang JK, Park IS. The changing patterns of liver abscess during the past 20 years--a study of 482 cases. Yonsei Med J. 1993 Dec;34(4):340-51. doi: 10.3349/ymj.1993.34.4.340. PMID 8128739